CLINICAL TRIAL: NCT03563950
Title: A Phase I, Open-Label Study to Evaluate the Effect of Rifampin on the Single Dose Pharmacokinetics, Safety and Tolerability of BMS-986224 in Healthy Subjects
Brief Title: An Investigational Study to Evaluate the Effect of Rifampin on the Singe Dose of Experimental Medication BMS-986224 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV016-008
Record Dates: First submitted 2018-06-11; First posted 2018-06-20 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rifampin + BMS-986224 (Experimental): Oral administration
  Interventions: Drug: Rifampin; Drug: BMS-986224

INTERVENTIONS:
Drug: Rifampin — Specified dose on specified days
Drug: BMS-986224 — Specified dose on specified days

SUMMARY:
The purpose of this study is to investigate if the blood levels of experimental medication BMS-986224 will be changed when given together with Rifampin, an antibiotic that affects specific enzymes involved with the breakdown of BMS-986224.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy participant, as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* Body mass index (BMI)of 18.0to 30.0 kg/m2, inclusive, at screening

Exclusion Criteria:

* Women of childbearing potential
* Any significant acute or chronic medical illness
* Current or recent (within 3 months of study treatment administration) gastrointestinal disease that could affect absorption or history of cholecystectomy

Other protocol defined inclusion/exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-986224 | 5 days
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] of BMS-986224 | 5 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of BMS-986224 | 5 days

SECONDARY OUTCOMES:
Biomarker plasma concentrations of BMS-986224 | 5 days
Time of maximum observed plasma concentration (Tmax) of BMS-986224 | 5 days
Terminal elimination half-life (T-HALF) of BMS-986224 | 5 days
Metabolite of BMS-986224 Cmax | 5 days
Metabolite of BMS-986224 AUC(0-T) | 5 days
Metabolite of BMS-986224 AUC(INF) | 5 days
Incidence of nonserious adverse events (AE) | 17 days
Incidence of serious adverse events (SAE) | 30 days
Incidence of AEs leading to discontinuation | 17 days
Composite results of vital signs, electrocardiograms, physical examinations,and clinical laboratory tests | 18 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PRA Health Sciences, Salt Lake City, Utah, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm